CLINICAL TRIAL: NCT01329770
Title: Phase II Double-blind Randomized Placebo-controlled 1-way Crossover Trial to Investigate Safety and Efficacy of the Ascorbic Acid and Tocopherol for the Treatment of the Fragile X Syndrome
Brief Title: Safety and Efficacy Study of Antioxidants for the Treatment of the Fragile X Syndrome
Acronym: SXF-TRA152
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yolanda de Diego Otero (Other)
Responsible Party: Sponsor-Investigator, Yolanda de Diego Otero, MSc PhD, The Mediterranean Institute for the Advance of Biotechnology and Health Research
Organization: The Mediterranean Institute for the Advance of Biotechnology and Health Research (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-017837-23
Record Dates: First submitted 2011-03-29; First posted 2011-04-06 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Fragile X Syndrome
Keywords: Neurodevelopmental disability; Hyperactivity; Anxiety; Cognitive problems; Behavioural symptoms; Fragile X syndrome; Autism; inherited Genetic condition
MeSH Terms: conditions — Fragile X Syndrome; Spasm; Anxiety Disorders; Behavioral Symptoms; Autistic Disorder | interventions — Ascorbic Acid; alpha-Tocopherol; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ascorbic Acid and alpha-tocopherol (Experimental): Two daily doses of the combination of antioxidants, administered at breakfast and dinner
  Interventions: Dietary Supplement: Ascorbic Acid (Vitamin C) and Alpha-tocopherol (Vitamin E)
- Placebo (Placebo Comparator): Two daily doses of placebo, administered at breakfast and dinner
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ascorbic Acid (Vitamin C) and Alpha-tocopherol (Vitamin E) — * Vitamin E (D-alpha-Tocopherol) 10 mg/kg/day (with a maximum of 600mg/day)
  * Vitamin C (L-Ascorbic Acid) 10 mg/kg/day (with a maximum of 800mg/day) For 12 weeks
  Arms: Ascorbic Acid and alpha-tocopherol
Dietary Supplement: Placebo — Two daily dose of placebo, administered at breakfast and dinner for 12 weeks
  Arms: Placebo

SUMMARY:
The Fragile X syndrome (FXS) was first described by Dr. Martin and Dr. Bell in 1943, in families with several patients affected by sex-linked mental disability. This disorder is the most common cause of inherited mental disability. The prevalence of the Fragile X syndrome has been established at 1 in 2,500 males and 1 in 4000 females.

Despite moderate to severe mental retardation, fragile X patients exhibit macroorchidism, an elongated face, long ears, connective tissue dysplasia, hyperactivity, autistic-like and stereotypical behaviours, speech delay and increased sensory sensitivity.

Objective: To evaluate the effect of the combination of the antioxidant Ascorbic acid and tocopherol, as therapy of the Fragile X Syndrome in young males.

Hypothesis: It is proposed that part of the pathophysiology of the central nervous system in the animal model of the fragile X syndrome may be determined by oxidative stress. In addition, Fragile X patients showed a significantly low level of ascorbic acid in plasma. The biochemical characteristics of oxidative stress may be reversed in the FMR1-KO mice, by a chronic treatment with antioxidant compounds such as tocopherol or melatonin, it may also normalize several hallmarks of the Syndrome such as hyperactivity, anxiety and cognitive deficits. The normalization of the oxidative stress is proposed as a new therapeutic pathway to alleviate conditions caused by an excess of free radicals that are crucial in neurodevelopmental diseases such as autism, down syndrome and other diseases of the central nervous system.

DETAILED DESCRIPTION:
* Objective: To evaluate the effect of the combination of the antioxidant Ascorbic acid and tocopherol, as therapy of the Fragile X Syndrome in young males.
* Design: Pilot clinical trial, Phase II , 6-month randomized, double-blind placebo-controlled one-way crossover clinical trial, with two treatment periods of 12 weeks duration.
* Setting: IMABIS Foundation. Carlos Haya Hospital, Malaga.
* Subjects: Children aged 5-11 years (infants) and 12-18 years (adolescents) diagnosed with Fragile X syndrome.
* Intervention: 30 participants randomly assigned, to receive antioxidant vitamins C (ascorbic acid) and vitamin E (d-alpha-tocopherol) once a day or placebo for 12 weeks double-blind. In Study Period 2, all participants receive (open) active treatment. Outcome measures: improvement in plasma antioxidant levels, oxidative stress (indicated by glutathione status, thiobarbituric acid reacting substances (TBARS) and carbonyl content of proteins) and HPA axis response. Behavioral problems will be studied using "Developmental behavior checklist" and "Teacher's and Parent´s Questionnaire, C. Keith Conners", also learning improvement will be analyzed using "Wechsler Intelligence Scale for children" at 0, 3, 6 months during the trial and 3 months after completing the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Molecular genetics diagnosis of the syndrome (number of CGG repeats in the FMR1 gene over 200).
* Presenting characteristic symptoms of fragile X syndrome.
* Patients older than 6 years and younger that 19 years.
* Signed informed consent by parents and/or legal tutor prior to enrolment in the trial.
* Both parents and patients must commit to participate for the duration of the 30 week trial.

Exclusion Criteria:

* The study excludes individuals with other neurological disorders not linked to the syndrome.
* Patients that have had serious medical problems in the previous 12 months.
* Are taking more than 100mg of vitamin E or vitamin C daily for the past 4 months.
* Have physical problems, mental or sensory impairments that preclude the assessment of effectiveness.
* Hypersensitivity to any component of the preparation.

Ages: 6 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes in the baseline Conner's Parent and Teacher Scales at 12 and 24 weeks | Baseline, week 12, week 24
  Hyperactivity scales: Conners Parent and Teacher Questionnaire, realized before starting treatment, 12 weeks and 24 weeks after beginning the treament.

SECONDARY OUTCOMES:
Change in the baseline measure of the Inventory of behaviour development (DBC-P24) at 12 and 24 weeks | Baseline, week 12 and week 24
  Inventory of behaviour development (DBC-P24) will be realized before starting, 12 weeks and 24 weeks after beginning the treatment
Wechsler Intelligence Scale for children | baseline, week 12 and week 24
  Wechsler Intelligence Scale for children will be used at base line and 12 weeks after beginning the treatment
Composite measure of blood and urine. | Baseline, week 12 and week 24
  Safety Evaluation through blood and urine measurement. The following studies will be done at base line, 12 and 24 weeks after beginning the treatment:
  1. Hematology
  2. Biochemical
  3. Determination of adrenal axis.
  4. Oxidative status.
  5. Analysis of urine density, pH, protein, glucose, ketone bodies, bilirubin, blood, nitrite, urobilinogen, leukocytes, urinary sediment, sodium, chlorine, potassium.

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda de Diego Otero, PhD, Principal Investigator — IMABIS Foundation. Hospital Carlos Haya. Malaga; Lucia M Perez Costillas, MD PhD, Principal Investigator — Hospital Carlos Haya. Malaga
Locations (1):
- Psychiatric Service. Hospital Carlos Haya, Málaga, Malaga, Spain

REFERENCES:
- [Background] de Diego-Otero Y, Romero-Zerbo Y, el Bekay R, Decara J, Sanchez L, Rodriguez-de Fonseca F, del Arco-Herrera I. Alpha-tocopherol protects against oxidative stress in the fragile X knockout mouse: an experimental therapeutic approach for the Fmr1 deficiency. Neuropsychopharmacology. 2009 Mar;34(4):1011-26. doi: 10.1038/npp.2008.152. Epub 2008 Oct 8. PMID 18843266
- [Background] Romero-Zerbo Y, Decara J, el Bekay R, Sanchez-Salido L, Del Arco-Herrera I, de Fonseca FR, de Diego-Otero Y. Protective effects of melatonin against oxidative stress in Fmr1 knockout mice: a therapeutic research model for the fragile X syndrome. J Pineal Res. 2009 Mar;46(2):224-34. doi: 10.1111/j.1600-079X.2008.00653.x. Epub 2008 Dec 23. PMID 19141086
- [Background] el Bekay R, Romero-Zerbo Y, Decara J, Sanchez-Salido L, Del Arco-Herrera I, Rodriguez-de Fonseca F, de Diego-Otero Y. Enhanced markers of oxidative stress, altered antioxidants and NADPH-oxidase activation in brains from Fragile X mental retardation 1-deficient mice, a pathological model for Fragile X syndrome. Eur J Neurosci. 2007 Dec;26(11):3169-80. doi: 10.1111/j.1460-9568.2007.05939.x. Epub 2007 Nov 14. PMID 18005058
- [Derived] de Diego-Otero Y, Calvo-Medina R, Quintero-Navarro C, Sanchez-Salido L, Garcia-Guirado F, del Arco-Herrera I, Fernandez-Carvajal I, Ferrando-Lucas T, Caballero-Andaluz R, Perez-Costillas L. A combination of ascorbic acid and alpha-tocopherol to test the effectiveness and safety in the fragile X syndrome: study protocol for a phase II, randomized, placebo-controlled trial. Trials. 2014 Sep 3;15:345. doi: 10.1186/1745-6215-15-345. PMID 25187257
- See also: Foundation IMABIS — http://www.imabis.org